CLINICAL TRIAL: NCT00323648
Title: Does it Make Sense to Give Postoperative Antibiotics to Patients With an Uncomplicated Acute Cholecystitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2006/111
Record Dates: First submitted 2006-05-07; First posted 2006-05-09 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2014-12

CONDITIONS: Uncomplicated Acute Cholecystitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- postoperatively antibiotics (Experimental)
  Interventions: Drug: Whether or not giving postoperatively antibiotics to patients with an uncomplicated acute cholecystitis

INTERVENTIONS:
Drug: Whether or not giving postoperatively antibiotics to patients with an uncomplicated acute cholecystitis — Whether or not giving postoperatively antibiotics to patients with an uncomplicated acute cholecystitis.

SUMMARY:
Each patient is preoperatively treated once profylactic with intraveneous antibiotics. Postoperatively, one group will be treated with intraveneous antibiotics during 5 days. The other group will receive no antibiotics.

ELIGIBILITY:
Inclusion Criteria:

* Uncomplicated acute cholecystitis < 5 days(confirmed by echography and blood sample)
* > 18 years old

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2006-05; Primary Completion 2010-05 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Postoperative complications (abces, infection of the wound) | day 2, day of discharge and dag 21

SECONDARY OUTCOMES:
Duration of hospitalisation | Day O to day of discharge

CONTACTS AND LOCATIONS:
Overall Officials: Frederik Berrevoet, MD, Principal Investigator — University Hospital, Ghent
Locations (2):
- University Hospital Ghent, Ghent, Belgium
- Hamad Medical Corporation, Doha, Qatar

REFERENCES:
- See also: Website of the University Hospital Ghent — http://www.uzgent.be